CLINICAL TRIAL: NCT02229266
Title: Randomised Controlled Phase-2 Trial to Determine the Efficacy of Adoptive Immunotherapy With Haploidentical Natural Killer Cells in High-risk Acute Myeloid Leukemia
Brief Title: Randomised Controlled Phase-2 Trial to Determine the Efficacy of Adoptive Immunotherapy With NK Cells in High-risk AML
Acronym: HINKL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-HINKL1-059
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; high-risk AML; acute myeloid leukemia; NK cells; haploidentical natural killer cells; immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NK cells (Experimental): Infusion of haploidentical NK cells after immunosuppression with cyclophosphamide and fludarabine, followed by immunostimulatory treatment with interleukin-2
  Interventions: Biological: NK cells
- Control Intervention (Active Comparator): 1 cycle of consolidation chemotherapy with high-dose cytarabine
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Biological: NK cells
  Other Names: CD3-negative/ CD56-positive NK cells from HLA-haploidentical family; donors
  Arms: NK cells
Drug: Cytarabine — 1 cycle of consolidation chemotherapy with high-dose cytarabine
  Other Names: chemotherapy
  Arms: Control Intervention

SUMMARY:
The trial investigates the efficacy of adoptive immunotherapy with haploidentical natural killer cells compared to standard chemotherapy (after first complete remission) in patients with a high-risk acute myeloid leukemia being older than 65 years of age and not eligible for allogeneic transplantation

DETAILED DESCRIPTION:
Randomised controlled phase-2 trial to determine the efficacy of adoptive immunotherapy with haploidentical natural killer cells in high-risk acute myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML other than acute promyelocytic leukemia (APL) according to WHO criteria
* In AML defined by cytogenetic aberrations the proportion of blasts may be <20%
* Age ≥60 years
* Clinical performance corresponding to ECOG score 0-2
* High-risk karyotype
* <5% myeloblasts in bone marrow ≥21 days after beginning of most recent chemotherapy
* maximal two preceding chemotherapy cycles
* Potentially available haploidentical family donor (child/ sibling), willing and fit for NK cell donation

Exclusion Criteria:

* AML with favorable or intermediate risk cytogenetic features
* Persistent aplasia following preceding chemotherapy
* Relapsed or refractory AML
* Known pre-existing autoimmune diseases
* Any severe concomitant condition which makes it undesirable for the patient to participate in the study
* Any condition which could jeorpadize compliance of the protocol
* Participation in another clinical trial during or within 4 weeks before study entry

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04-22 (Actual); Study Completion 2017-04-22 (Actual)

PRIMARY OUTCOMES:
2-year overall survival | 2 years after study inclusion
  measure time of survival of each patiente up to 2 years after study inclusion

SECONDARY OUTCOMES:
Time to relapse | 2 years after study inclusion
  evaluate time to relapse for 2 years after study inclusion for each patient; calculate cumulative incidence of relapse
Relapse-free survival | 2 years after study inclusion
Yield and purity of NK cells (CD3-CD56+) after CD3 depletion and CD56 enrichment | timepoint of application of NK cells
NK cell analysis | 2 years after study inclusion
Clinical performance (ECOG score) | 2 years after study inclusion
Incidence and severity of GVHD | 6 months after start of treatment
Incidence of (S)AEs | 5 weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bornhäuser, Prof. Dr. med., Principal Investigator — Universitätsklinikum Dresden
Locations (3):
- Germany (3):
  - Klinikum Bayreuth, Bayreuth
  - Klinikum Chemnitz, Chemnitz
  - Universitätsklinikum Dresden, Dresden

REFERENCES:
- See also: Study Alliance Leukemia — http://www.sal-aml.org
- See also: Universitätsklinikum Dresden, Medizinische Klinik I — http://www.uniklinikum-dresden.de/das-klinikum/kliniken-polikliniken-institute/mk1